CLINICAL TRIAL: NCT06133660
Title: Influence of Intravitreal Aqueous Tamponade on Lens Status and Ocular
Status: Completed | Type: Observational
Sponsor: Bo Jia (Other)
Responsible Party: Sponsor-Investigator, Bo Jia, M.D., Second Hospital of Jilin University
Organization: Second Hospital of Jilin University (Other)
Other Study IDs: second hospital of JilinU
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Aqueous Tamponade; Cataract
Keywords: aqueous tamponade; cataract; lens thickness; axial length; pars plana vitrectomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPV（pars plana vitrectomy） group
  Interventions: Procedure: pars plana vitrectomy
- Silicone oil removal group
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Procedure: pars plana vitrectomy — pars plana vitrectomy and Silicone oil removal to distinguish subjects
  Other Names: Silicone oil removal

SUMMARY:
To observe the effects of vitreous cavity Balanced salt solution (BSS) tamponade on the state of the lens and related parameters of the eye, and whether the changes of the above parameters are correlated with age, gender, diabetes or not, etc., so as to provide references for the diagnosis and treatment of related diseases and scientific research.

ELIGIBILITY:
Inclusion Criteria:

* ① Patients undergoing vitrectomy for diabetic retinopathy, epiretinal membranes, macular hole, retinal detachment, and other diseases;

  * Patients who underwent vitreous silicone oil tamponade and vitreous silicone oil removal due to various causes; ③ Intraoperative BSS was used for fill the vitreous cavity; ④ Before treatment, inform the patient that the clinical data may be used in clinical research, and the patient and his family are informed and sign the informed consent.

Exclusion Criteria:

* ① The operation eye was intraocular lens or cataract extraction during operation; ② Suspensory ligament relaxation or rupture, ciliary body detachment or transaction, lens dislocation, endophthalmitis, traumatic cataract;

  * intraoperative lens injury; ④ patients who refused to participate in the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergoing vitrectomy for diabetic retinopathy, epiretinal membranes, macular hole, retinal detachment, and other diseases, or underwent vitreous silicone oil tamponade and vitreous silicone oil removal due to various causes
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
degree of lens opacity | 1 year
lens thickness | 1 year

SECONDARY OUTCOMES:
anterior chamber depth | 1 year
axial length | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: Yes